CLINICAL TRIAL: NCT00575094
Title: A Phase 3, Multicenter, Open-label Study Evaluating the Safety and Efficacy of Intravenous Tigecycline to Treat Hospitalized Japanese Subjects With Community-acquired Pneumonia
Brief Title: Study Evaluating the Safety and Efficacy of Intravenous Tigecycline to Treat Hospitalized Japanese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3074A1-3331
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2009-05-27 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-06

CONDITIONS: Community-Acquired Infections
MeSH Terms: conditions — Community-Acquired Infections | interventions — Tigecycline

INTERVENTIONS:
Drug: tigecycline — Dosage form: Tigecycline 50 mg for injection (Lyophilized powder in 5 mL vial) Dosage frequency: Tigecycline 100 mg loading followed by 50 mg every 12 hrs (bid) Duration of therapy: 7 to 14 days

SUMMARY:
To purpose of this study is to assess the safety and tolerability of intravenous (IV) tigecycline in hospitalized subjects of Japanese descent with community-acquired pneumonia (CAP).

DETAILED DESCRIPTION:
This is a multicenter, open-label study evaluating the safety and efficacy of tigecycline in the treatment of Japanese subjects with CAP. Subjects with clinical signs and symptoms of CAP who meet the eligibility requirements will be considered for enrollment. Qualifying subjects will be assigned to receive tigecycline via IV administration for 7 to 14 consecutive days. The exact duration of administration of the study drug will be at the discretion of the investigator, based on the subject's condition. Subjects will be followed for safety until the test-of-cure (TOC) assessment 10 to 21 days after the last dose of therapy, and for efficacy until TOC assessment.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized Japanese descent subjects known or suspected to have CAP with a severity that requires IV antibiotic treatment.
* Chest radiograph within 48 hours before the first dose of IV test article showing the presence of a new infiltrate.
* The presence of fever or hypothermia within 24 hours before the first administration of test article, and of at least two signs/symptoms of CAP within 24 hours before the first administration of test article.

Exclusion Criteria:

* Any concomitant condition that, in the opinion of the investigator, would preclude an evaluation of a response or make it unlikely that the contemplated course of therapy could be completed.
* Hospital-acquired pneumonia, other lung disease including viral, fungal, or parasitic pneumonia, immunosuppressive conditions, and other illness, which affect evaluation of safety and efficacy of tigecycline.
* Known or suspected hypersensitivity to tigecycline or tetracyclines, or contraindication for these antibiotics.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (8):
- Japan (8):
  - Toyota-shi, Aichi-ken
  - Kurume-shi, Fukuoka
  - Yanagawa-shi, Fukuoka
  - Asahikawa-shi, Hokkaido
  - Funaishikawa, Ibaraki
  - Yokohama, Kanagawa
  - Suwa-shi, Nagano
  - Kiyose-shi, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in Japan from November 2007 to February 2008.
Pre-assignment Details: Subjects were screened up to 24 hours.
Groups:
- Tigecycline: Intravenous (IV) administration for 7 to 14 consecutive days at the discretion of the investigator.
Period: Overall Study
Arm/Group | Tigecycline
Started | 9
Completed | 6
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tigecycline
Number analyzed (Participants) | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 62.78 (18.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients by Clinical Response at Test-of-Cure (TOC) Visit.
Description: Clinical response: Cure=all initial signs/symptoms of pneumonia (SSx) improved; chest x-ray (CXR)improved/stable; no other antibiotics for pneumonia; no worsening or new SSx. Failure=persistence or worsening SSx; no clinical improvement or initial improvement with clinically important worsening; other antimicrobials for pneumonia CXR progression; death > study day 2 due to pneumonia. Indeterminate=unable to determine outcome for nonstudy drug/infection reasons (eg, lost to follow-up); death ≤2 days after first dose for any reason, or >2 days but before TOC visit for non-pneumonia reason.
Time Frame: 8 weeks
Population: All patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tigecycline
Number analyzed (Participants) | 9
participants
  Cure | 6
  Failure | 2
  Indeterminate | 1

ADVERSE EVENTS:
Arm/Group | Tigecycline
Serious Adverse Events (participants affected / at risk) | 1
Other Adverse Events (participants affected / at risk) | 9
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Tigecycline
Liver Dysfunction (Hepatobiliary disorders) | 1/9
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Tigecycline
Diarrhea (Gastrointestinal disorders) | 4/9
Nausea (Gastrointestinal disorders) | 9/9
Stomach Disorder (Gastrointestinal disorders) | 1/9
Vomiting (Gastrointestinal disorders) | 4/9
Alanine aminotransferase increased (Investigations) | 1/9
Aspartate aminotransferase increased (Investigations) | 1/9
Bilirubin conjugated increased (Investigations) | 1/9
Blood bilirubin increased (Investigations) | 1/9
Blood urea increased (Investigations) | 1/9
Anorexia (Metabolism and nutrition disorders) | 1/9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1/9
Headache (Nervous system disorders) | 1/9
Insomnia (Psychiatric disorders) | 1/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.